CLINICAL TRIAL: NCT05110872
Title: COMET Study 2: Effects of Cigarette and E-cigarette Flavor Restrictions on Cigarette Demand and Substitution in the Experimental Tobacco Marketplace
Brief Title: Cigarette and E-cigarette Flavors Manipulations in the Experimental Tobacco Marketplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VT IRB# 20-827; P01CA217806 (NIH)
Record Dates: First submitted 2021-10-11; First posted 2021-11-08 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Use Disorder
Keywords: Cigarette; E-cigarette; Behavioral Economics; Tobacco Control
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Intervention Model Description: Participants will complete different purchasing scenarios in the Experimental Tobacco Marketplace in which different cigarette and e-cigarette flavors are available. In all scenarios, a range of other tobacco products will also be available.
Who Masked: Investigator
Masking Description: The study design included automated randomization of the conditions per person at the time of completion, via Qualtrics Software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol cigarette smokers (Experimental): Adults (21 y.o. and older) who smoke ate least 10 menthol cigarettes per day will be recruited.
  Interventions: Behavioral: Cigarette flavor restricted and e-cigarette flavor restricted; Behavioral: Cigarette flavor restricted and e-cigarette flavor unrestricted; Behavioral: Cigarette flavor unrestricted and e-cigarette flavor restricted; Behavioral: Cigarette flavor unrestricted and e-cigarette flavor unrestricted
- Non-menthol cigarette smokers (Experimental): Adults (21 y.o. and older) who smoke ate least 10 non-menthol cigarettes per day will be recruited.
  Interventions: Behavioral: Cigarette flavor restricted and e-cigarette flavor restricted; Behavioral: Cigarette flavor restricted and e-cigarette flavor unrestricted; Behavioral: Cigarette flavor unrestricted and e-cigarette flavor restricted; Behavioral: Cigarette flavor unrestricted and e-cigarette flavor unrestricted

INTERVENTIONS:
Behavioral: Cigarette flavor restricted and e-cigarette flavor restricted — 1. Tobacco cigarettes will be available in the Experimental Tobacco Marketplace
  2. Tobacco-flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
Behavioral: Cigarette flavor restricted and e-cigarette flavor unrestricted — 1. Tobacco cigarettes will be available in the Experimental Tobacco Marketplace
  2. Tobacco-flavored and a range of flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
Behavioral: Cigarette flavor unrestricted and e-cigarette flavor restricted — 1. Tobacco and menthol cigarettes will be available in the Experimental Tobacco Marketplace
  2. Tobacco-flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
Behavioral: Cigarette flavor unrestricted and e-cigarette flavor unrestricted — 1. Tobacco and menthol cigarettes will be available in the Experimental Tobacco Marketplace
  2. Tobacco-flavored and a range of flavored e-cigarettes will be available in the Experimental Tobacco Marketplace

SUMMARY:
This is a one-session study that participants complete remotely including consent, Experimental Tobacco Marketplace purchases, and assessments to examine the effects of cigarette and e-cigarette flavors on cigarette demand and substitution in the Experimental Tobacco Marketplace.

DETAILED DESCRIPTION:
This study uses a mixed design (within-subject repeated measures and between-group). Participants will be assigned to two different groups according to their preferred cigarette flavor (tobacco/menthol). Every participant will complete behavioral tasks and make hypothetical purchases of tobacco products in an online store under four different scenarios: a) e-cigarette flavor restricted and cigarette flavor restricted, b) e-cigarette flavor unrestricted and cigarette flavor restricted, c) e-cigarette flavor restricted and cigarette flavor unrestricted, d) e-cigarette flavor unrestricted and cigarette flavor unrestricted.

ELIGIBILITY:
Inclusion Criteria:

* currently smoke at least 10 cigarettes per day
* have smoked at least 100 cigarettes (lifetime), and
* are 21 years of age or older.

Exclusion Criteria:

* inaccurate identification of usual brand of cigarette's as menthol or non-menthol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Menthol Cigarette Smokers: Adults (21 y.o. and older) who smoke ate least 10 menthol cigarettes per day will be recruited.
  Cigarette flavor restricted and e-cigarette flavor restricted: 1) Tobacco cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
  Cigarette flavor restricted and e-cigarette flavor unrestricted: 1) Tobacco cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored and a range of flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
  Cigarette flavor unrestricted and e-cigarette flavor restricted: 1) Tobacco and menthol cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
  Cigarette flavor unrestricted and e-cigarette flavor unrestricted: 1) Tobacco and menthol cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored and a range of flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
- Non-menthol Cigarette Smokers: Adults (21 y.o. and older) who smoke ate least 10 non-menthol cigarettes per day will be recruited.
  Cigarette flavor restricted and e-cigarette flavor restricted: 1) Tobacco cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
  Cigarette flavor restricted and e-cigarette flavor unrestricted: 1) Tobacco cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored and a range of flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
  Cigarette flavor unrestricted and e-cigarette flavor restricted: 1) Tobacco and menthol cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
  Cigarette flavor unrestricted and e-cigarette flavor unrestricted: 1) Tobacco and menthol cigarettes will be available in the Experimental Tobacco Marketplace 2) Tobacco-flavored and a range of flavored e-cigarettes will be available in the Experimental Tobacco Marketplace
Period: Overall Study
Arm/Group | Menthol Cigarette Smokers | Non-menthol Cigarette Smokers
Started | 140 | 162
Completed | 140 | 162
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menthol Cigarette Smokers | Non-menthol Cigarette Smokers | Total
Number analyzed (Participants) | 130 | 133 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.15 (13.31) | 49.77 (13.95) | 49.46 (13.63)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 70 | 58 | 128
  Male | 60 | 75 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 15 | 35
  Not Hispanic or Latino | 110 | 118 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 2 | 14
  White | 112 | 124 | 236
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 130 | 133 | 263
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 19.79 (13.05) | 18.18 (8.82) | 18.99 (10.94)

OUTCOME MEASURES:

1. Primary Outcome: Spent the Budget on E-cigarettes for Each Condition
Description: Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Product availability in the ETM depended on the experimental condition. The average percentage of budget spent on e-cigarettes as a function of the restriction of cigarettes and/or e-cigarettes will be assessed.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of spent budget
Arm/Group | Menthol Cigarette Smokers | Non-menthol Cigarette Smokers
Number analyzed (Participants) | 130 | 133
percentage of spent budget
  Cigarette and E-cigarette Restriction | 10.64 (1.36) | 14.87 (1.44)
  Cigarette Restriction | 14.74 (1.62) | 14.65 (1.38)
  E-cigarette restriction | 8.20 (1.17) | 15.03 (1.42)
  No Restriction on Cigarettes or E-cigarettes | 11.35 (1.45) | 16.07 (1.47)

2. Primary Outcome: Spent Budget on Cigarettes for Each Condition
Description: Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Product availability in the ETM depended on the experimental condition. The average percentage of the budget spent on cigarettes as a function of the restriction of cigarettes and/or e-cigarettes will be assessed.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of spent budget
Arm/Group | Menthol Cigarette Smokers | Non-menthol Cigarette Smokers
Number analyzed (Participants) | 130 | 133
percentage of spent budget
  Cigarette and E-cigarette Restriction | 55.04 (2.56) | 65.82 (2.03)
  Cigarette Restriction | 53.05 (2.57) | 65.80 (2.02)
  E-cigarette Restriction | 73.60 (2.13) | 65.72 (2.00)
  No Restriction on Cigarettes or E-cigarettes | 72.05 (2.14) | 65.20 (2.03)

ADVERSE EVENTS:
Time Frame: approximately 19 days
Arm/Group | Menthol Cigarette Smokers | Non-menthol Cigarette Smokers
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/162
Other Adverse Events (participants affected / at risk) | 0/140 | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT05110872/Prot_SAP_ICF_000.pdf